CLINICAL TRIAL: NCT01618851
Title: Phase II Study to Evaluate the Efficacy of Intensity Modulated Radiation Therapy With Hypofractionated Radiosurgical Boosts in the Treatment of Clinically Localized Prostate Cancer
Brief Title: Phase II Study to Evaluate Conventional Radiation Therapy Followed by Radiosurgical Boost in Clinically Localized Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Sean Collins, M.D., PhD, Assistant Professor, Georgetown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 2009-599
Record Dates: First submitted 2012-06-12; First posted 2012-06-13 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMRT with SBRT Boost (Experimental): Patients with clinically localized prostate cancer will be treated with three radiosurgical treatments (6.5 Gy per fraction to PTV) followed by IMRT (45 Gy in 25 fractions) over 6-7 weeks.
  Interventions: Radiation: Radiotherapy with IMRT and CyberKnife Boost

INTERVENTIONS:
Radiation: Radiotherapy with IMRT and CyberKnife Boost — Inverse planning using the CyberKnife planning system will be employed. The treatment plan used for each treatment will be based on an analysis of the volumetric dose including dose-volume histogram (DVH) analyses of the PTV and critical normal structures. The homogeneous CT model shall be used.
  The prescribed PTV dose of 19.5 Gy shall be given in 3 fractions using the CyberKnife. At least three fiducials should be identified for each treatment. If fewer than three fiducials can be tracked, then additional fiducials will be placed, and the patient replanned. Fiducial locations in the images will be extracted and compared to the fiducial locations in the CT scans to estimate target movements.
  For IMRT, Daily doses of 180 cGy are to be delivered to the PTV 5 days a week to a total dose of 4500 cGy in 25 fractions.

SUMMARY:
This phase II study designed to prospectively evaluate the efficacy and morbidity of IMRT with CyberKnife radiosurgical boosts for clinically localized prostate cancer. Patients will be treated with three radiosurgical treatments (6.5 Gy per fraction) followed by IMRT (45 Gy in 25 fractions).

DETAILED DESCRIPTION:
This is a phase II study designed to prospectively evaluate the efficacy and morbidity of IMRT with CyberKnife radiosurgical boosts for clinically localized prostate cancer. Patients with clinically localized prostate cancer will be treated with three radiosurgical treatments (6.5 Gy per fraction to the PTV) followed by IMRT (45 Gy in 25 fractions). Treatment will be completed over a 6-7 week period.

The hypothesis is that for patients with clinically localized adenocarcinoma of the prostate, CyberKnife Radiosurgery delivered to the prostate is efficacious with acceptable toxicity in combination with IMRT.

Subjects will have toxicity evaluation and AUA score on the last day of treatment. At 1 month following treatment, subjects will be assessed for acute toxicity and will fill out AUA form, SF-12, EPIC-26, SHIM and Utilization of Sexual Rx/Devices. At 3, 6, 12, 18 and 24 month intervals (and every 6 months thereafter, through year 5, and annually through year 10, if investigators opt to continue past year 5), subjects will be seen and evaluated, including a history, physical exam, performance status, PSA, toxicity evaluation, and AUA score. In addition, at 6 months, 12 months and annually thereafter, the SF-12, EPIC-26, SHIM and Utilization of Sexual Medications/Devices will be administered. A prostate biopsy will be performed at time of biochemical or local clinical failure, and is encouraged at 2 years following treatment and at time of distant failure. A bone scan will be performed at the time of biochemical failure, or when the subject develops signs of symptoms suggesting metastatic disease.

Acute side effects (≤ 90 days of treatment start) will be assessed using the NCI Toxicity Criteria version 3.0.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate (Biopsy within one year of enrollment)
* Signed Study-Specific COnsent
* PSA within 60 days of registration
* Baseline AUA score is less than 20

Exclusion Criteria:

* Prior Pelvic radiotherapy
* Prior Radical Prostate surgery
* Recent (within 5 years) or concurrent cancers other than non-melanoma skin cancer
* Medical or psychiatric illness that would interfere with treatment or follow-up
* Implanted hardware adjacent to the prostate that would prohibit appropriate treatment planning and/or treatment delivery.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-11; Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Local failure | 2 years after radiotherapy.
  To estimate the rate of local failure as assessed by 2 year post-radiotherapy prostate biopsies. (Studies with the CyberKnife radiosurgery would be worthwhile for prostate cancer patients if the rate of local control was > 70%)

SECONDARY OUTCOMES:
Gastrointestinal and genitourinary toxicity | During 5 years following the CyberKnife SRS treatment for prostate cancer
  To estimate the proportion of patients who develop late grade 3-5 gastrointestinal and genitourinary toxicity observed during the five years following CyberKnife SRS for prostate cancer.
Biochemical disease-free survival (bDFS) | 2 years after radiotherapy
  To assess secondary efficacy endpoints: Biochemical disease-free survival (bDFS) assessed using both Phoenix and ASTRO definitions, disease-free survival, disease-specific survival, time to failure, overall survival, duration of local control, and proportion of distant failure at 2 years.
Patient Reported Quality of Life: American Urological Association symptom index | During the 5 years following radiotherapy
  American Urological Association (AUA) symptom index to assess bothersome urinary symptoms on a scale of 0-5 (0 = not at all, 5 = almost always) for assessment. Numbers are tallied and total score of 1-7 MILD, 8-19 MODERATE, 20-35 SEVERE. Patient reported quality of life is recorded as; 0-6 (0=no symptoms, 6=extremely unhappy).
Patient Reported Quality of Life: Expanded Prostate Cancer Index Composite-26 (EPIC-26) | During the 5 years following radiotherapy
  Expanded Prostate Cancer Index Composite-26 contains 26 questions assessing: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal therapy. Response range 0-4 (0 =no problem, 4=big problem).
Patient Reported Quality of Life: Sexual Health Inventory for Men (SHIM) | During the 5 years following radiotherapy
  Sexual Health Inventor for Men Sexual health classifies severity of erectile dysfunction with the following breakpoints: 1-7 Severe ED 8-11 Moderate ED 12-16 Mild to Moderate ED 17-21 Mild ED
Patient Reported Quality of Life: Utilization of Sexual Medications and Devices | During the 5 years following radiotherapy
  Utilization of Sexual Medications/Devices is optional and assesses the use of erectile aids by patients treated for prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Collins, MD,PhD, Principal Investigator — Georgetown University Hospital

REFERENCES:
- [Derived] Dess RT, Devasia TP, Aghdam N, Jackson WC, Soni PD, Smith CP, Mitchell AL, Suy S, Hamstra DA, Jolly S, Nguyen PL, Feng FY, Schipper MJ, Skolarus TA, Miller DC, Wittmann DA, Collins SP, Spratt DE. Patient-Reported Sexual Aid Utilization and Efficacy After Radiation Therapy for Localized Prostate Cancer. Int J Radiat Oncol Biol Phys. 2018 Jun 1;101(2):376-386. doi: 10.1016/j.ijrobp.2018.01.055. Epub 2018 Jan 31. PMID 29487023